CLINICAL TRIAL: NCT00831610
Title: Post-bariatric Abdominoplasty: Skin Sensation Evaluation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodolpho Alberto Bussolaro, MD. PhD., Doctor, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UNIFESP-712/06
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Obesity; Hypesthesia
Keywords: bariatric surgery; plastic surgery; abdominal wall; skin; sensation; abdominoplasty
MeSH Terms: conditions — Obesity; Hypesthesia | interventions — Bariatric Surgery; Gastric Bypass; Abdominoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STUDY (Other): 1. Female healthy volunteers (25 to 55 years old) with normal weight.
  2. Morbid Obese women waiting for bariatric surgery.
  3. Post-bariatric female patients, 25 to 55 years old, MORE than 12 months of weight stability, pendular abdominal wall, clinical conditions to anchor-line abdominoplasty without flap undermining. Skin Evaluation before the abdominoplasty.
  4. Group 3, submitted to anchor-line abdominoplasty without flap undermining.
  Interventions: Procedure: Bariatric surgery (Roux-en-Y Gastric Bypass) + Post-bariatric abdominoplasty.; Procedure: Roux-en-Y gastric bypass (bariatric surgery) + Post-bariatric abdominoplasty (without flap undermining)
- CONTROL (Other): Group 3: Post-bariatric female patients, 25 to 55 years old, LESS than 12 months of weight stability, pendular abdominal wall, clinical conditions to anchor-line abdominoplasty without flap undermining. Who will be submitted to abdominoplasty after the study period.
  Interventions: Procedure: Roux-en-Y gastric bypass (bariatric surgery) + Post-bariatric abdominoplasty (without flap undermining)

INTERVENTIONS:
Procedure: Bariatric surgery (Roux-en-Y Gastric Bypass) + Post-bariatric abdominoplasty. — Surgical removal of the exceeding skin and adiposity of the abdominal wall by one midline vertical fuse and one supra-pubic horizontal fuse. Skin suture without flap undermining and with low tension.
  Other Names: Anchor-line abdominoplasty; Abdominoplasty; Post-bariatric plastic surgery
  Arms: STUDY
Procedure: Roux-en-Y gastric bypass (bariatric surgery) + Post-bariatric abdominoplasty (without flap undermining) — Bariatric surgery Plastic surgery Abdominoplasty

SUMMARY:
The purpose of this study is to quantify the skin sensation of the anterior abdominal wall of the post-bariatric patients submitted to anchor-line abdominoplasty without flap undermining.

Additional purposes were: quantify topographically the abdominal skin sensation of the Normal weight, Morbid Obese and Former Morbid Obese after bariatric surgery (before and after the abdominoplasty - excess skin surgical removal without flap undermining -> Anchor Line Abdominoplasty).

DETAILED DESCRIPTION:
Abdominoplasty performed in post-bariatric patients presents more post-operative complications than in non post-bariatric patients. Surgical techniques that provokes less complications are required.

Anchor-line abdominoplasty is a technique published in the years 1950 as well the first bariatric proceedings. Abdominoplasty without flap undermining is feasible in pendular abdominal wall of the former morbidly obese women with scarred abdomen.

Classical abdominoplasty (with flap undermining) is known to impair significantly the skin sensation. Post-bariatric abdominoplasty without flap undermining keeps the skin sensation unaltered since the early post-operative period.

Now that the post-bariatric anchor-line abdominoplasty improves the abdominal wall contour by removing the exceeding, pendular and striated skin saving the perforant skin sensory nerves. Could this technique improve the skin sensation of the anterior abdominal wall of the post-bariatric patients?

ELIGIBILITY:
Inclusion Criteria:

* Former morbidly obese women with Body Mass Index superior of 40kg/m2.
* Post-bariatric surgery: Roux en Y gastric bypass.
* Clinical conditions to perform a plastic surgery.

Exclusion Criteria:

* Diabetes.
* Peripheral neuropathy.
* Deny to sign the Informed Consent Term.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Innocuous static tactile sensation in grams per square millimeters (g/mm2) by nylon monofilaments aesthesiometer. | Day before the surgical intervention and 6th month after for Study group.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolpho A Bussolaro, PhD fellow, Principal Investigator — Federal University of São Paulo; Elvio B Garcia, Professor, Study Chair — Federal University of São Paulo; Lydia M Ferreira, Chairwoman, Study Director — Federal Universtity of São Paulo
Locations (1):
- Federal Universtiy of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Bussolaro RA, Garcia EB, Barbosa MV, Omonte IR, Huijsmans JP, Bariani RL, Ferreira LM. Post-bariatric abdominoplasty: skin sensation evaluation. Obes Surg. 2010 Jul;20(7):855-60. doi: 10.1007/s11695-008-9747-9. Epub 2008 Nov 4. PMID 18982397
- See also: Institutional ethics committee web-site. — http://www.unifesp.br/reitoria/orgaos/comites/etica/index.php